CLINICAL TRIAL: NCT01699373
Title: A Randomised Controlled Trial on Ultrasound-assisted Spinal Anaesthesia
Brief Title: A Trial on Ultrasound-assisted Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UGSA/2010
Record Dates: First submitted 2012-09-30; First posted 2012-10-03 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-02

CONDITIONS: Spinal Anaesthesia; Ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound-assisted (Experimental): Pre-procedural ultrasound scan performed
  Interventions: Procedure: Ultrasound scan
- Manual Palpation (No Intervention)

INTERVENTIONS:
Procedure: Ultrasound scan — Pre-procedural ultrasound scan was performed
  Arms: Ultrasound-assisted

SUMMARY:
A randomised controlled trial comparing the use of pre-procedural ultrasound scanning with manual palpation to identify landmarks for performance of spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* undergoing surgery amenable to spinal anaesthesia

Exclusion Criteria:

* Patient refusal
* contraindications to regional anaesthesia
* known allergy to local anaesthetics
* bleeding diathesis
* inability to provide informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2011-April 2012 Changi General Hospital
Period: Overall Study
Arm/Group | Ultrasound-assisted | Manual Palpation
Started | 85 | 85
Completed | 85 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound-assisted | Manual Palpation | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 85 | 170
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 61.1 (13.3) | 63.7 (12.6) | 62.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 45 | 75
  Male | 55 | 40 | 95
Region of Enrollment [Number; unit: participants]
  Singapore | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of First-attempt of Spinal Anaesthesia
Time Frame: During procedure
Measure: Number; unit: participants
Arm/Group | Ultrasound-assisted | Manual Palpation
Number analyzed (Participants) | 85 | 85
participants | 54 | 44

2. Secondary Outcome: Time Taken to Perform Spinal Anaesthesia
Time Frame: During procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ultrasound-assisted | Manual Palpation
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Baseline characteristics not equal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes